CLINICAL TRIAL: NCT05731804
Title: A Multicenter, Non-randomized, Open-label, Parallel Controlled Phase I Clinical Study to Evaluate the Pharmacokinetics, Safety and Tolerability of SIM0417/Ritonavir After a Single Dose in Subjects With Renal or Hepatic Impairment
Brief Title: Hepatic Impairment and Renal Impairment Study of SIM0417 Combined With Ritonavir
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIM0417-105
Record Dates: First submitted 2023-01-18; First posted 2023-02-16 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Renal Impairment; Hepatic Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 of Part A (Experimental): Subjects with mild renal impairment(SIM0417 600 mg; Ritonavir100 mg )
  Interventions: Drug: SIM0417 600 mg; Ritonavir100 mg
- Cohort 2 of Part A (Experimental): Subjects with moderate renal impairment(SIM0417 375 mg; Ritonavir100 mg )
  Interventions: Drug: SIM0417 375 mg; Ritonavir100 mg
- Cohort 3 of Part A (Experimental): Subjects with normal renal function(SIM0417 600 mg; Ritonavir100 mg )
  Interventions: Drug: SIM0417 600 mg; Ritonavir100 mg
- Cohort 4 of Part A (Experimental): Subjects with normal renal function(SIM0417 375 mg; Ritonavir100 mg )
  Interventions: Drug: SIM0417 375 mg; Ritonavir100 mg
- Cohort 5 of Part B (Experimental): Subjects with moderate hepatic impairment (SIM0417 750 mg; Ritonavir100 mg )
  Interventions: Drug: SIM0417 750 mg; Ritonavir100 mg
- Cohort 6 of Part B (Experimental): Subjects with normal hepatic function(SIM0417 750 mg; Ritonavir100 mg )
  Interventions: Drug: SIM0417 750 mg; Ritonavir100 mg

INTERVENTIONS:
Drug: SIM0417 600 mg; Ritonavir100 mg — SIM0417 is single dosed, and ritonavir is administered 12 hours before SIM0417 administration (-12 hours), at the time of SIM0417 administration (0 hour), 12 hours (12 hours) after SIM0417 administration, and 24 hours (24 hours) after SIM0417 administration.
  Arms: Cohort 1 of Part A; Cohort 3 of Part A
Drug: SIM0417 375 mg; Ritonavir100 mg — SIM0417 is single dosed, and ritonavir is administered 12 hours before SIM0417 administration (-12 hours), at the time of SIM0417 administration (0 hour), 12 hours (12 hours) after SIM0417 administration, and 24 hours (24 hours) after SIM0417 administration.
  Arms: Cohort 2 of Part A; Cohort 4 of Part A
Drug: SIM0417 750 mg; Ritonavir100 mg — SIM0417 is single dosed, and ritonavir is administered 12 hours before SIM0417 administration (-12 hours), at the time of SIM0417 administration (0 hour), 12 hours (12 hours) after SIM0417 administration, and 24 hours (24 hours) after SIM0417 administration.
  Arms: Cohort 5 of Part B; Cohort 6 of Part B

SUMMARY:
This is a multicenter, nonrandomized, open-label, parallel controlled Phase I clinical study to evaluate the Pharmacokinetics, Safety and Tolerability of SIM0417 combined with ritonavir after a single dose in subjects with mild and moderate renal impairment, moderate hepatic impairment, normal renal function, and normal hepatic function. It is divided into Part A (subjects with mild/moderate renal impairment and subjects with normal renal function) and Part B (subjects with moderate hepatic impairment and subjects with normal hepatic function).

DETAILED DESCRIPTION:
This is a multicenter, non-randomized, open-label, parallel controlled Phase I clinical study to evaluate the Pharmacokinetics, Safety and Tolerability of SIM0417 combined with ritonavir after a single dose in subjects with mild and moderate renal impairment, moderate hepatic impairment, normal renal function, and normal hepatic function.

Part A includes 4 cohorts, each of which plans to enroll 6-12 subjects, for a total of 24-48 subjects. Participants will be allocated into normal renal function or mild/moderate renal impairment groups based on their estimated glomerular filtration rate.

Part B includes 2 cohorts, each of which plans to enroll 6-12 subjects, for a total of 12-24 subjects. Participants will be allocated into normal hepatic function or moderate hepatic impairment groups based on their Child-Pugh score.

Each subject will receive SIM0417 combined with ritonavir administration. SIM0417 is single-dosed, and ritonavir is administered 12 hours before SIM0417 administration (-12 hours), at the time of SIM0417 administration (0 hour), 12 hours (12 hours) after SIM0417 administration, and 24 hours (24 hours) after SIM0417 administration.

ELIGIBILITY:
Inclusion Criteria:

* ● PartA:

  * All subjects

    1. Fully understand the study content, process, and potential risks of this trial, and voluntarily sign the informed consent.
    2. Male and female subjects aged ≥18 years and ≤75 years old.
    3. Male subjects weigh ≥50 kg, female subjects weigh ≥45 kg; BMI ≥ 18 and ≤ 28 kg/m^2.
    4. The results of screening and baseline blood pregnancy examination of women of childbearing potential are negative, and they are willing to take effective contraceptive measures during the trial and within 3 months after the last administration of the investigational product, or have postmenopause or surgical sterilization; male subjects have no fertility plan during the trial and within 3 months after the last administration of the investigational product and voluntarily take effective contraceptive measures or have surgical sterilization.
  * Subjects with renal impairment

    1. Glomerular filtration rate should meet the following criteria ( eGFR = eGFR（CKD-EPI）× BSA / 1.73): Mild renal impairment ( CKD2 ) 60-89 mL/min (both values included; Moderate renal impairment ( CKD3 ) 30-59 mL/min (both values included).
    2. The renal function status is stable, and the GFR results of the two tests before administration (at least 3 days interval ) must be in the same CKD stage.
    3. No medication within 14 days before enrollment, or with a stable medication regimen for the treatment of renal impairment or other comorbidities (the type, dose or frequency of medication has not been adjusted for at least 2 weeks).
    4. Total bilirubin, ALT and AST ≤ 2 ×ULN.
    5. Be in acceptable physical condition except for renal impairment and complications, according to medical history inquiry, physical examination, vital signs, laboratory tests (Hematology, blood biochemistry, urinalysis, coagulation function, thyroid function ), 12-lead ECG, chest radiograph, thyroid ultrasound, abdominal ultrasound(judged by the investigator).
  * Subjects with normal renal function

    1. Age-matched (±10 years), weight-matched (±15kg), and gender-matched with subjects in the renal impairment group.
    2. Glomerular filtration rate( eGFR = eGFR（CKD-EPI）× BSA / 1.73)≥ 90 mL / min.
    3. Vital signs, physical examination, laboratory tests (Hematology, blood biochemistry, urinalysis, coagulation function, thyroid function ), 12 lead ECG, chest radiograph, abdominal ultrasound, thyroid ultrasound examination are normal or abnormal with no clinical significance.
* ● PartB

  * All subjects

    1. Fully understand the study content, process, and potential risks of this trial, and voluntarily sign the informed consent.
    2. Male and female subjects aged ≥18 years and ≤75 years old.
    3. Male subjects weigh ≥50 kg, female subjects weigh ≥45 kg; BMI ≥ 18 and ≤ 28 kg/m^2.
    4. The results of screening and baseline blood pregnancy examination of women of childbearing potential are negative, and they are willing to take effective contraceptive measures during the trial and within 3 months after the last administration of the investigational product, or have postmenopause or surgical sterilization; male subjects have no fertility plan during the trial and within 3 months after the last administration of the investigational product and voluntarily take effective contraceptive measures or have surgical sterilization.
  * Subjects with hepatic impairment

    1. With chronic ( diagnosis ≥ 6 months, stable disease ≥ 4 weeks ) moderate liver dysfunction ( Child-Pugh score: 7-9 points ) caused by viral hepatitis, alcoholic liver disease, autoimmune hepatitis, primary biliary cirrhosis or other causes ( except drug-induced liver injury ). If it is impossible to judge whether the disease is stable or not, 2 examinations must be carried out during the screening period with an interval of at least 2 weeks to judge the stable disease state. The investigators diagnosed chronic liver function damage according to standard diagnosis and treatment methods, combined with the subject's previous medical history, laboratory tests, liver biopsy or imaging examination and other documents, and then evaluated according to Child-Pugh classification (according to encephalopathy grade, ascites, serum albumin, serum bilirubin, prothrombin time prolongation in seconds).
    2. No medication within 14 days before enrollment, or with a stable medication regimen for the treatment of hepatic impairment or other comorbidities (the type, dose or frequency of medication has not been adjusted for at least 2 weeks).
    3. Glomerular filtration rate ( absolute eGFR = eGFR（CKD-EPI） × BSA / 1.73 ) ≥60 mL / min.
    4. Be in acceptable physical condition except for hepatic impairment and complications, according to medical history inquiry, physical examination, vital signs, laboratory tests (Hematology, blood biochemistry, urinalysis, coagulation function, thyroid function ), 12-lead ECG, chest radiograph, thyroid ultrasound, abdominal ultrasound(judged by the investigator).
  * Subjects with normal hepatic function

    1. Age-matched (±10 years), weight-matched (±15kg), and gender-matched with subjects in the hepatic impairment group.
    2. Total bilirubin, ALT and AST ≤ the upper limit of normal.
    3. Vital signs, physical examination, laboratory examination (Hematology, blood biochemistry, urinalysis, coagulation function, thyroid function ), 12-lead ECG, chest radiograph, abdominal ultrasound, thyroid ultrasound examination are normal or abnormal with no clinical significance.

Exclusion Criteria:

* ● PartA:

  * All subjects

    1. Breastfeeding women.
    2. Those with allergies, including a history of severe drug allergy or drug allergy; or may be allergic to the study drug or any excipients of the study drug.
    3. Difficulties in venous blood collection.
    4. With severe infection, trauma, major surgical operation, digestive system surgery, and affecting drug absorption within 4 weeks before screening.
    5. Within six months before screening, patients with myocardial infarction, severe/unstable angina pectoris, symptomatic congestive heart failure ( NYHA II-IV ), or history of supraventricular or ventricular arrhythmia or left ventricular impairment which was Clinically significant and requiring treatment or intervention.
    6. Participated in clinical trials of any drug intervention within 3 months before screening.
    7. Blood donation ≥ 400 mL within 3 months before screening, or received blood transfusion or blood products within 1 month before the screening.
    8. Those who are addicted to smoking or drinking within 3 months before screening, and who cannot stop smoking and drinking during the test, or those who have a positive breath test for alcohol. (Remarks: addicted to Smoking is defined as ≥5 cigarettes/day; alcoholism is defined as daily drinking exceeding the following standard amounts: 570 mL of beer, 750 mL of light beer, 200 mL of red wine or 60 mL of white wine, each containing about 20 g of alcohol ).
    9. With Drug abuse history or a positive drug abuse screen.
    10. Used any CYP3A4 potent inducer within 28 days before the first administration.
    11. Special diets ( including pitayas, mangoes, grapefruit, caffeine-containing foods or drinks, etc. ) or intense exercise were taken within 48 hours before the first administration of the study drug.
    12. Those who have been vaccinated within 1 month before screening (except for the COVID-19 vaccine), or who plan to be vaccinated during treatment / within 2 weeks after the last dose of study drug.
    13. 12-lead ECG at screening, QT interval (QTcF) corrected by Fridericia formula ≥ 470 msec (female)/450 msec (male).
    14. Be positive in SARS-CoV-2 nucleic acid test or SARS-CoV-2 antigen at screening.
    15. The investigator judges that there are other factors of subjects that are not suitable for participating in this trial.
  * Subjects with renal impairment

    1. Renal transplantation.
    2. Requires renal dialysis during the study.
    3. Urinary incontinence or anuria.
    4. In addition to the disease itself causing the diagnosis of renal impairment, subjects suffering from acute diseases of any other organs, and suffering any chronic diseases that may affect the in vivo process of the study drug (e.g.hepatic impairment, etc.)are inappropriate for participation in this trial(judged by the investigator).
    5. Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5×ULN), or significant clinically significant bleeding symptoms or definite hemorrhagic tendency within 3 months before screening, such as alimentary tract hemorrhage, gastric ulcer bleeding, etc., or are receiving thrombolytic anticoagulation therapy.
    6. At screening, systolic pressure >160 mmHg, diastolic pressure >100 mmHg; pulse >100 bpm.
    7. Combined virus infection ( anti-HCV positive, anti-HIV positive, HBsAg positive ) or syphilis infection.
  * Subjects with normal renal function

    1. WIth a history of cardiovascular, liver, kidney, digestive tract, immune, blood, endocrine, metabolism, cancer, mental and neurological diseases at the time of screening.
    2. At screening, systolic pressure <90 mmHg or >140 mmHg, diastolic pressure <60 mmHg or >90 mmHg; pulse <55 bpm or >100 bpm.
    3. Combined virus infection ( anti-HCV positive, anti-HIV positive, HBsAg positive ) or syphilis infection.
    4. Prescription, non-prescription and traditional Chinese medicine ( Chinese herbal medicine, Chinese patent medicine ) were used within 2 weeks before screening.
* ● PartB:

  * All subjects

    1. Breastfeeding women.
    2. Those with allergies, including a history of severe drug allergy or drug allergy; or may be allergic to the study drug or any excipients of the study drug.
    3. Difficulties in venous blood collection.
    4. With severe infection, trauma, major surgical operation, digestive system surgery, and affecting drug absorption within 4 weeks before screening.
    5. With six months before screening, patients with myocardial infarction, severe/unstable angina pectoris, symptomatic congestive heart failure ( NYHA II-IV ), or intervention of supraventricular or ventricular arrhythmia or left ventricular dysfunction, have clinical significance and require treatment.
    6. Participated in clinical trials of any drug intervention within 3 months before screening.
    7. Blood donation ≥ 400 mL within the first 3 months before screening, or received blood transfusion or blood products within 1 month before the screening.
    8. With addicted to smoking and drinking within 3 months before screening, cannot smoke or drink alcohol during the study period, or have a positive alcohol breath test. (Remarks: Smoking is defined as ≥5 cigarettes/day; alcoholism is defined as daily drinking exceeding the following standard amounts: 570 mL of beer, 750 mL of light beer, 200 mL of red wine or 60 mL of white wine, each containing about 20 g of alcohol ).
    9. With Drug abuse history or a positive drug abuse screen.
    10. Used any CYP3A4 potent inducer within 28 days before the first administration.
    11. Special diets ( including pitayas, mangoes, grapefruit, caffeine-containing foods or drinks, etc. ) or intense exercise were taken within 48 hours before the first administration of the study drug.
    12. Vaccines ( other than new coronavirus vaccines ) have been vaccinated within 1 month before screening or plan to be vaccinated during treatment or within 2 weeks after the last administration of the study drug.

        13.12-lead ECG at screening, QT interval (QTcF) corrected by Fridericia formula ≥ 470 msec (female)/450 msec (male).

    14. Be positive in SARS-CoV-2 nucleic acid test or SARS-CoV-2 antigen at screening.

    15. Other factors of subjects that are not suitable for participating in this trial(judged by the investigator).
  * Subjects with hepatic impairment

    1. Have ever received a liver transplant.
    2. With liver failure or with severe complications of cirrhosis.
    3. Patients with hepatic encephalopathy ( grade 3-4 hepatic encephalopathy according to Child-Pugh score ).
    4. Fluctuating or rapidly worsening liver function, manifested by extensive changes or deterioration of clinical symptoms and/or laboratory tests of liver damage symptoms during screening ( such as advanced ascites, fever, and active gastrointestinal bleeding ).
    5. Severe portal hypertension, or transjugular intrahepatic portosystemic shunt, or esophageal variceal bleeding in the past 2 months.
    6. Suspected or diagnosed with liver cancer or other malignant tumors.
    7. Received drugs with clear potential hepatotoxicity (such as halothane, etc.) within 3 months before administration of study.
    8. In addition to the disease itself causing the diagnosis of hepatic impairment, subjects suffering from acute diseases of any other organs, and any chronic diseases that may affect the in vivo process of the study drug (e.g.renal impairment, etc.) are inappropriate for participation in this trial(judged by the investigator).
    9. Anticoagulant therapy with warfarin or related coumarins.
    10. At screening, systolic pressure >160 mmHg, diastolic pressure >100 mmHg; pulse >100 bpm.
    11. Combined virus infection ( anti-HIV positive ) or syphilis infection.
  * Subjects with normal hepatic function

    1. WIth a history of cardiovascular, liver, kidney, digestive tract, immune, blood, endocrine, metabolism, cancer, mental and neurological diseases at the time of screening.
    2. At screening, systolic pressure <90 mmHg or >140 mmHg, diastolic pressure <60 mmHg or >90 mmHg; pulse <55 bpm or >100 bpm.
    3. Combined virus infection ( anti-HCV positive, anti-HIV positive, HBsAg positive ) or syphilis infection.
    4. Prescription, non-prescription and traditional Chinese medicine ( Chinese herbal medicine, Chinese patent medicine ) were used within 2 weeks before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cmax of SIM0417 in Part A | Up to 48 hours from SIM0417 administration
  Cmax of SIM0417 in Part A when SIM0417 combined with ritonavir
AUC0-t of SIM0417 in Part A | Up to 48 hours from SIM0417 administration
  AUC0-t of SIM0417 in Part A when SIM0417 combined with ritonavir
AUC0-∞ of SIM0417 in Part A | Up to 48 hours from SIM0417 administration
  AUC0-∞ of SIM0417 in Part A when SIM0417 combined with ritonavir
Cmax of SIM0417 in Part B | Up to 48 hours from SIM0417 administration
  Cmax of SIM0417 in Part B when SIM0417 combined with ritonavir
AUC0-t of SIM0417 in Part B | Up to 48 hours from SIM0417 administration
  AUC0-t of SIM0417 in Part B when SIM0417 combined with ritonavir
AUC0-∞ of SIM0417 in Part B | Up to 48 hours from SIM0417 administration
  AUC0-∞ of SIM0417 in Part B when SIM0417 combined with ritonavir

SECONDARY OUTCOMES:
Tmax of SIM0417 in Part A | Up to 48 hours from SIM0417 administration
  Tmax of SIM0417 in Part A when SIM0417 combined with ritonavir
t1/2 of SIM0417 in Part A | Up to 48 hours from SIM0417 administration
  t1/2 of SIM0417 in Part A when SIM0417 combined with ritonavir
CL/F of SIM0417 in Part A | Up to 48 hours from SIM0417 administration
  CL/F of SIM0417 in Part A when SIM0417 combined with ritonavir
Vz/F of SIM0417 in Part A | Up to 48 hours from SIM0417 administration
  Vz/F of SIM0417 in Part A when SIM0417 combined with ritonavir
Ae of SIM0417 in Part A | Up to 96 hours from SIM0417 administration
  Ae of SIM0417 in Part A when SIM0417 combined with ritonavir
protein binding of SIM0417 in Part A | Up to 12 hours from SIM0417 administration
  Plasma protein binding rate of SIM0417 in Part A when SIM0417 combined with ritonavir
Vital Signs in Part A | Up to 5 days from the start of administration
  Number of Participants With Clinically Notable Vital Signs in Part A
ECG in Part A | Up to 5 days from the start of administration
  Number of Participants With Clinically Notable Electrocardiogram (ECG) Values in Part A
Laboratory Tests in Part A | Up to 5 days from the start of administration
  Number of Participants With Clinically Notable Laboratory Tests in Part A
Adverse Events in Part A | Up to 14 days from the start of administration
  Number of Participants With Adverse Events in Part A
Tmax of SIM0417 in Part B | Up to 48 hours from SIM0417 administration
  Tmax of SIM0417 in Part B when SIM0417 combined with ritonavir
t1/2 of SIM0417 in Part B | Up to 48 hours from SIM0417 administration
  t1/2 of SIM0417 in Part B when SIM0417 combined with ritonavir
CL/F of SIM0417 in Part B | Up to 48 hours from SIM0417 administration
  CL/F of SIM0417 in Part B when SIM0417 combined with ritonavir
Vz/F of SIM0417 in Part B | Up to 48 hours from SIM0417 administration
  Vz/F of SIM0417 in Part B when SIM0417 combined with ritonavir
Protein binding of SIM0417 in Part B | Up to 12 hours from SIM0417 administration
  Plasma protein binding rate of SIM0417 in Part B when SIM0417 combined with ritonavir
Vital Signs in Part B | Up to 5 days from the start of administration
  Number of Participants With Clinically Notable Vital Signs in Part B
ECG in Part B | Up to 5 days from the start of administration
  Number of Participants With Clinically Notable Electrocardiogram (ECG) Values in Part B
Laboratory Tests in Part B | Up to 5 days from the start of administration
  Number of Participants With Clinically Notable Laboratory Tests in Part B
Adverse Events in Part B | Up to 14 days from the start of administration
  Number of Participants With Adverse Events in Part B

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Principal Investigator — Shandong First Medical University
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No